CLINICAL TRIAL: NCT04320641
Title: The Effect of Acupressure and Yoga on Premenstrual Symptoms and Quality of Life in Coping With PMS
Brief Title: The Effect of Acupressure and Yoga on Premenstrual Symptoms and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Didem Kucukkelepce, Didem Kucukkelepce, Adiyaman University Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Inonu Universty
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Premenstrual Syndrome; Nursing Caries
Keywords: PMS,; YOGA; NURSING; HEALTH QUALITY
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Acupressure; Yoga

STUDY DESIGN:
Who Masked: Participant
Masking Description: * who do not have regular periods (between 21-35 days),
  * Has a psychiatric diagnosis,
  * Having any gynecological disease (anornal uterine bleeding, fibroids, ovarian cyst etc.)
  * Using contraceptive drugs,
  * With tissue deformity in its extremities, Any health problems that may prevent physical exercise
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- acupressure (Experimental)
  Interventions: Other: ACUPRESSURE
- music (Experimental)
  Interventions: Other: ACUPRESSURE
- control (No Intervention)

INTERVENTIONS:
Other: ACUPRESSURE — Acupressure points were determined in a certain order considering the direction of the meridian. The order of application was in the form of Spleen 6th point (SP 6) and 4 point of the Large Intestine (Li 4). In total, 4 points in the upper / lower extremities and 6 acupressure points along with parallel points were studied in each attempt.
  Other Names: YOGA
  Arms: acupressure; music

SUMMARY:
The research was carried out to determine the effect of acupressure and yoga applied to cope with PMS on premenstrual symptoms and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* have regular menstrual cycle

Exclusion Criteria:

* Has a psychiatric diagnosis,

  * Having any gynecological disease (anornal uterine bleeding, fibroids, ovarian cyst etc.)
  * Using contraceptive drugs,
  * With tissue deformity in its extremities, Any health problems that may prevent physical exercise

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
premenstrual syndrome scale | 12 weeks
WHOQOL-BREF-TR | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Didem Simsek Kucukkelepce, Adi̇yaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No